CLINICAL TRIAL: NCT00005839
Title: A Phase I Study of Oxaliplatin in Combination With Capecitabine in Metastatic/Recurrent Solid Tumors
Brief Title: Oxaliplatin Plus Capecitabine in Treating Patients With Metastatic or Recurrent Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067854; U01CA062505 (NIH); CHNMC-PHI-25; CHNMC-IRB-99130; NCI-T99-0005
Record Dates: First submitted 2000-06-02; First posted 2003-04-21 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Capecitabine; Oxaliplatin

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of oxaliplatin combined with capecitabine in treating patients who have metastatic or recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of capecitabine when administered in combination with oxaliplatin in patients with metastatic or recurrent solid tumors. II. Determine the toxicities of this treatment regimen in this patient population.

OUTLINE: This is a dose escalation study of capecitabine. Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed for disease progression and survival.

PROJECTED ACCRUAL: A total of 12-15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic or recurrent solid tumor that has failed standard therapy or for which no standard therapy exists No known brain metastases or carcinomatosis meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Karnofsky 60-100% Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 times normal AST no greater than 2.5 times normal Renal: Creatinine normal OR Creatinine clearance greater than 60 mL/min Calcium no greater than 12 mg/dL Cardiovascular: No symptomatic congestive heart failure No unstable angina pectoris No cardiac arrhythmia Other: No evidence of neuropathy No history of allergies to platinum compounds or antiemetics that would preclude study No other uncontrolled illness (e.g., ongoing or active infection) No medical, social, or psychological factors that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas) and recovered Prior fluorouracil or cisplatin allowed Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Recovered from prior surgery Other: At least 30 days since prior investigational drugs No concurrent antiretroviral therapy (HAART)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Study Chair — University of Southern California
Locations (3):
- United States (3):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California